CLINICAL TRIAL: NCT06291805
Title: Phenotyping and Characterization of Danish Wild-type Transthyretin Amyloidosis Cardiomyopathy Patients: A Cross-sectional Study
Brief Title: Phenotyping and Characterization of wtATTR-CM (TRACE 1)
Status: Recruiting | Type: Observational
Sponsor: Steen Hvitfeldt Poulsen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, DMSc., Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Other Study IDs: 1-10-72-189-23
Record Dates: First submitted 2024-01-30; First posted 2024-03-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Transthyretin Amyloidosis; Transthyretin Amyloid Cardiomyopathy; Wild-Type Transthyretin-Related (ATTR)Amyloidosis; Quality of Life
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blod and endomyocardial biopsies. No DNA test are made.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- wtATTR-CM patients (n = 100): Clinical history, physical examination, ECG, advanced echocardiography, blood and urine samples, cardiac magnetic resonance imaging (CMRI), and QoL questionaires (KCCQ, EQ-5Q-5L and ATTR-QoL)).
  Subgroup with these patient (n = 10): A endomyocardial biopsy.
- Control (n = 20): Blood and urine samples. To rule out cardiac disease: clinical history, physical examination, ECG and advanced echocardiography.

SUMMARY:
Descriptive cross-sectional study on 100 consecutive ATTRwt-CM patients reflecting all NAC stages aiming primarily to investigate ATTRwt-CM patient's quality of life (QoL) measures and their relation to ATTRwt-CM severity. Secondarily aiming to investigate the possibility to measure misTTR and fragTTR in plasma and urine and to detect fragTTR in endomyocardial biopsies from ATTRwt-CM patients. To investigate whether misTTR and fragTTR levels are correlated with ATTRwt-CM severity.

DETAILED DESCRIPTION:
Hypothesis:

1. We hypothesize that more severe wild-type amyloidosis cardiomyopathy (ATTRwt-CM) according to clinical, biochemical, and diagnostic imaging parameters are correlated with worse quality of life (QoL) for patients.
2. We expect misfolded (misTTR) and/or fragmented transthyretin (fragTTR) to be measurable in plasma and/or urine and fragTTR to be detectable in endomyocardial biopsies from patients with ATTRwt-CM. We expect the values of misTTR and fragTTR to be correlated with the severity of ATTRwt-CM according to clinical, biochemical, and diagnostic imaging parameters. We expect the level of fragTTR from endomyocardial biopsies to be correlated with plasma levels of fragTTR.

Method:

ATTRwt-CM patients: Prospective inclusion of 100 consecutive ATTRwt-CM patients reflecting all NAC stages (40 patients from NAC disease stage 1, 40 patients from NAC disease stage II and 20 patients from NAC disease stage III). Patients will be recruited from the out-patient amyloidosis clinic at Aarhus University hospital. Patients will be thoroughly clinically assessed.

Control patients:

A control cohort of 20 age- and gender-matched heart-healthy patients will be included for comparison of total/mis-/fragTTR values.

The investigating into QoL, bio markers and the analyses on cardiac MR imaging markers will hopefully provide us with tools to evaluate and monitor disease progression and response to treatment.

ELIGIBILITY:
Group 1: wtATTR-CM patients

Inclusion Criteria:

* Patients > 18 years diagnosed with ATTRwt-CM by:
* endomyocardial biopsy
* DPD scintigraphy with Perugini grade 2-3 where variant amyloidosis is ruled out due to genetic testing.
* Informed oral and written consent

Exclusion Criteria:

* AL amyloidosis (light-chain amyloidosis).
* Myelomatosis
* Waldenström macroglobulinemia

Group 2: Control group

Inclusion Criteria:

* Patients > 18 years
* Informed oral and written consent

Exclusion Criteria:

* Known cardiovascular disease including ischemic heart disease, heart failure, atrial fibrillation, presence of a pacemaker, or malignant hypertension. Well-controlled hypertension is acceptable.
* Suspicion of cardiac amyloidosis assessed through clinical history, physical examination, ECG, and echocardiography focusing on "red flags":
* Echocardiography with:
* Myocardial hypertrophy (septum >11 mm)
* Apical sparing in LV-GLS
* Infiltrative changes in the right ventricle free wall, thickened atrioventricular valves, or thickened atrial septum
* Symptoms of polyneuropathy
* Low voltage on ECG or discrepancy between left ventricular thickness and ECG amplitude indicative of low voltage
* Atrioventricular block (AV block)
* Bilateral carpal tunnel syndrome
* Surgery for spinal stenosis
* Elevated troponin I or NT-pro-BNP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Including variating severity of wtATTR-CM by including 40 patients with NAC stage 1, 40 patients with NAC stage 2, and 20 patients with NAC stage 3. Furthermore, including a healthy control group in order to examine normal values of mis- and frag-TTR
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Investigation of cardiac amyloidosis severity in patients with Wild-type Transthyretin Amyloidosis Cardiomyopathy. | Through study completion, 2 years.
  Amyloid severity will be addressed using primarily NAC-stages and NYHA-class. Furthermore, we will use NT-pro-BNP, findings on echo (stroke volume, ejectionfraction and global longitudional strain) and finding on CMRI (LV mass, T1 myocardial values and extracellular volume).
Investigation of the relations between cardiac amyloid severity and patient quality of life in patients with Wild-type Transthyretin Amyloidosis Cardiomyopathy. | Through study completion, 2 years.
  Quality of life will be addressed using KCCQ summary score, EQ-5D Utility score and VAS ranging score and ATTR-QOL total score.
Assessment of transthyretin and pathogenic fragments and relation to cardiac amyloid severity in patients with Wild-type Transthyretin Amyloidosis Cardiomyopathy | Through study completion, 2 years.
  Transthyretin (TTR) will be measured as follows: total TTR, misfolded TTR and fragmented TTR in plasma and misfolded TTR and fragmented TTR in urine.

SECONDARY OUTCOMES:
Validation of a new amyloid specific questionnaire (ATTR-QoL) in comparison with Kansas City Cardiomyopathy Questionnaire (KCCQ) | Through study completion, 2 years.
  Comparing ATTR-QOL total score to KCCQ summary score and EQ-5D Utility score and VAS ranging score.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Arrhus N, Denmark

IPD SHARING:
Plan to Share IPD: No